CLINICAL TRIAL: NCT05314764
Title: Population Pharmacokinetics of Cefiderocol During Acute Pulmonary Exacerbations in Adult Patients With Cystic Fibrosis
Brief Title: Cefiderocol Pharmacokinetics in Adult Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Shionogi Inc. (Industry); Keystone Bioanalytical, Inc. (Unknown); Indiana University Health Methodist Hospital (Other); University of Pittsburgh Medical Center (Other); University of Texas (Other)
Responsible Party: Principal Investigator, Joseph L. Kuti, PharmD, Associate Director, CAIRD, Hartford Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HHC-2022-0078
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis; Pneumonia, Bacterial
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia, Bacterial | interventions — Cefiderocol

STUDY DESIGN:
Intervention Model Description: Open-label, descriptive, pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cefiderocol (Experimental): Participants will receive intravenous cefiderocol at a dosing regimen consistent with the current prescribing information and according estimated renal function. Each dose will be infused over 3 hours.
  Interventions: Drug: Cefiderocol

INTERVENTIONS:
Drug: Cefiderocol — Patients will receive intravenous cefiderocol every 6 to 8 hours for 4 to 6 doses.
  Other Names: Fetroja

SUMMARY:
There is established evidence that adult patients with Cystic Fibrosis (CF) may have altered antibiotic pharmacokinetics compared with non-CF patients. Cefiderocol is a newly approved broad spectrum intravenous siderophore cephalosporin antibiotic, which has potent in vitro activity against multidrug resistant Pseudomonas aeruginosa, Burkholderia cepacia complex, Achromobacter species, and Stenotrophomonas maltophilia, all pathogens implicated in CF pulmonary exacerbations. This study will determine the pharmacokinetics and tolerability of cefiderocol in 12 adult CF patients admitted for a pulmonary exacerbation at one of 4 participating hospitals in the US. Patients will remain on standard of care IV antibiotics and receive 4-6 doses of cefiderocol 2 grams infused over 3 hours every 6-8 hours, depending on kidney function. Blood will be sampled after the final dose to determine concentrations and pharmacokinetics of cefiderocol. Safety and tolerability will be assessed throughout the 2 day study.

DETAILED DESCRIPTION:
Participants will receive 4-6 doses of cefiderocol 2 grams every 6-8 hours, in addition to standard intravenous antibiotic therapy selected by the site. Just prior and then after the final dose, a total of nine blood samples will be collected to measure cefiderocol concentrations. Data will be fit to a population pharmacokinetic model. The final model will be utilized in a Monte Carlo simulation to determine the probability of several different dosing regimens retaining concentrations above the minimum inhibitory concentration (MIC) for at least 75% of the dosing interval. These data will be utilized to determine an optimized dosing regimen for adults with CF.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF
* Acute pulmonary exacerbation as the primary reason for admission to the hospital with requirement to receive systemic antibiotic treatment

Exclusion Criteria:

* Females that are pregnant and/or breastfeeding
* History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic (a history of mild rash to a cephalosporin followed by uneventful re-exposure is not a contraindication)
* History of a lung transplant at any time in the past or any other organ transplantation (e.g., liver) within the last 6 months
* Moderate to severe renal dysfunction defined as a creatinine clearance < 60 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight) or requirement for continuous renal replacement therapy or hemodialysis
* A hemoglobin less than 8 gm/dL at baseline
* Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Clearance | 0, 1.5, 3, 3.25, 4, 5, 6, and 8 hours after the final dose
  This outcome determines the clearance of cefiderocol over the dosing interval.
Volume of Distribution | 0, 1.5, 3, 3.25, 4, 5, 6, and 8 hours after the final dose
  This outcome determines the volume of distribution of cefiderocol over the dosing interval.

SECONDARY OUTCOMES:
Probability of Target Attainment at 4 mcg/mL | 24 hours
  This simulated outcome indicates the likelihood that cefiderocol will retain drug concentrations above the MIC for >/= 75% of the dosing interval at an MIC of 4 mcg/ml when administered as a 2g every 8 hour dose infused over 3 hour in patients up to a creatinine clearance of 120 ml/min. This analysis is conducted via a Monte Carlo simulation using the population pharmacokinetic parameter estimates and dispersion from the 12 participants who contributed pharmacokinetic data to the study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Kuti, PharmD, Principal Investigator — Hartford Hospital
Locations (4):
- United States (4):
  - Hartford Hospital, Hartford, Connecticut
  - IU Health University Hospital, Indianapolis, Indiana
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Clements University Hospital, Dallas, Texas